CLINICAL TRIAL: NCT06187259
Title: Efficacy of Smart Burs II ® in Selective Caries Removal in Permanent Molars: Randomized Controlled Trial
Brief Title: Comparative Study Between Smart Bur II and Traditional Carbide Bur in Selective Removal of Caries in Permanent Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Caries removal by polymer burs
Record Dates: First submitted 2023-11-29; First posted 2024-01-02 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2023-11

CONDITIONS: Dental Caries in Children

STUDY DESIGN:
Who Masked: Participant
Masking Description: single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- carbide bur group (Active Comparator): carbide burs are extremely hard and can withstand high temperatures. Because of their hardness, carbide burs can maintain a sharp cutting edge and can be used many times without becoming dull. They are best operated at high speeds with light pressure.
  Carbide dental bur was designed to, efficiently, remove non-decalcified enamel and dentin, yet, it does not facilitate the differentiation between carious and normal dentin, during cavity preparation.
  Interventions: Device: caries removal by carbide bur
- polymer bur II group (Experimental): Polymer bur tools resemble conventional burs in appearance, but they are made of unique polymer material rather than metal. The cutting edges are not spiral, like those of a shovel. The polymer material was designed to be softer than healthy dentin (Knoop hardness 70-90) but harder than carious, softening dentin (Knoop hardness 50-70) (Knoop hardness 0-30). Therefore, it has a knoop hardness of 50 kg/mm2, and its cutting elements effectively remove soft dentin but cannot remove healthy dentin.
  Interventions: Device: caries removal by polymer bur II

INTERVENTIONS:
Device: caries removal by carbide bur — caries was removed using a slow-speed handpiece and round carbide burs in sizes #12, #14, and #16, based on the lesion's size. When hard dentin was found using a dental probe, carious dentin removal was stopped.
  Arms: carbide bur group
Device: caries removal by polymer bur II — carious tissue was removed utilizing smart polymer burs of sizes #4, #6, and #8, depending on the cavity's size, running at a slow speed without water coolant, in circular motions from the center of the lesion outward. Carious dentin removal ceased when the instrument became macroscopically abraded and sharpened and could no longer remove tooth tissues.
  Arms: polymer bur II group

SUMMARY:
A more biological and conservative technique of caries removal has emerged with minimally invasive restorative dentistry's advent. As a result, Smart Burs II has become a self-limiting, sensitive tool for removing caries. The current study aimed to validate and contrast the polymer burs' efficacy (Smart Burs II) versus conventional burs (Carbide burs) for infected carious dentin's selective removal in permanent first molars. Thirty permanent first molars fulfilling the inclusion criteria were chosen in 8-11 years old children with class I occlusal carious lesions. Group 1 (n=15) and Group 2 (n=15) were randomly assigned to have carious dentin removed utilizing standard carbide bur and a smart Bur II, consecutively. By employing caries detector dye, the effectiveness of caries removal was quantified as 0, 1, 2, 3, 4, or 5. The volume of removed carious tissue was recorded using impression material which was inserted into a calibrated insulin syringe. A statistically significant difference was discovered in the volume of removed carious tissue between both groups, while the efficiency of caries removal using either bur has no significant difference. Smart Bur II was more conservative in the carious dentin's removal than carbide bur. Smart Bur II was as efficient as carbide bur in caries removal.

DETAILED DESCRIPTION:
One of the prime goals of the evolution of minimally invasive dentistry is conserving healthy tooth structure by eliminating infected carious dentin while retaining impacted carious dentin intact and minimizing the needless destruction of teeth. Dentin carious lesions is formed of two distinct layers that differ from one another regarding their microscopic structure and physiological and bacteriological characteristics. The external superficial infected layer is soft, heavily contaminated by bacterial invasion, and incapable of being repaired owing to the collagen fibers' irreversible denaturation. While the affected dentin, which is a hard substance with few bacteria and can be remineralized due to limited collagen degradation, is located beneath the infected layer.

Conventional caries removal could possibly be traumatic as it tends to remove both infected and affected dentin, which may induce an unneeded weakening of the tooth structure and often leads to overextended cavities. Moreover, it has deleterious thermal influences on the pulp. Accordingly, the dental industry has recently witnessed the emergence of the polymer bur, which manufacturers claim is the best for selectively removing caries while minimizing the patient's discomfort. By introducing a polymer prototype bur in 2003, a potential substitute for traditional techniques of removing carious dentin has emerged. This self-limiting polymer bur is known as SmartBurTM, a variant of SmartPrepTM (SS White, Lakewood, NJ, USA). It is a single-use bur-like instrument constructed of a polymer with a lower hardness than healthy dentin. Different sizes are available; #4, #6, and #8 for right angle latch handpieces.

Polymer bur tools resemble conventional burs in appearance, but they are made of unique polymer material rather than metal. The cutting edges are not spiral, like those of a shovel. The polymer material was designed to be softer than healthy dentin (Knoop hardness 70-90) but harder than carious, softening dentin (Knoop hardness 50-70) (Knoop hardness 0-30). Therefore, it has a knoop hardness of 50 kg/mm2, and its cutting elements effectively remove soft dentin but cannot remove healthy dentin.

Materials and methods Sample size calculation The minimum required sample size will be 15 molars in each group. Thus, a total of thirty permanent first molars will be divided into two groups for this study. The sample size was computed as per G*Power software version 3.1.9.3.

Allocation of samples A 1:1 allocation ratio was used to allocate each of the 30 selected permanent first molars to either Group 1 (Carbide Bur group) or Group 2 (Smart Bur II group).

Clinical Procedures and Grouping At the beginning of the dental visit, the "tell-show-do" method was performed, in which the child was introduced to all instruments and equipment used in the treatment session14. A periapical radiograph was taken for each carious molar. The proper isolation was conducted for the selected molars using a rubber dam and suction. local anesthesia was administered during the trial for each patient. The volume of the unprepared carious cavity, for both groups, was measured using impression material (Zhermack Oranwash L light c-silicone), which was inserted in a calibrated insulin syringe and consequently injected into the cavity before caries removal.

After recording the cavity's volume , the impression material was washed with water. The outline form of the cavity of all selected molars was established using a high-speed handpiece and round carbide bur. The removal of carious lesions was carried out for all the selected carious teeth, and they were split into two groups, as per the types of burs used for the removal of caries:

Carbide bur group (Group 1):

Using a slow-speed handpiece and round carbide burs in sizes #12, #14, and #16, based on the lesion's size, caries was removed. When hard dentin was found using a dental probe, carious dentin removal was stopped.

Smart Bur II group (Group 2):

As per the manufacturer's recommendations, carious tissue was removed utilizing smart polymer burs of sizes #4, #6, and #8, depending on the cavity's size, running at a slow speed without water coolant, in circular motions from the center of the lesion outward. Carious dentin removal ceased when the instrument became macroscopically abraded and sharpened and could no longer remove tooth tissues.

Caries detector dye (Red Detector, Cerkamed, Medical Company, Poland) was applied to all treated teeth of both groups as one drop on the defective area and waited 5-10 seconds. After that, irrigation with water for ten seconds was applied as recommended by the manufacturer's instructions. After drying the cavity, the examination was executed using the dental mirror to detect stained dentin sites. Points intensively dyed in red indicated residual caries. Then, the stained dentin was selectively removed by carbide and polymer burs according to each group. This process was frequent until no stain persisted in the cavity. After the full removal of caries in both groups, the cavity volume was again recorded using the same previous procedures of cavity volume measurements.

Assessment procedures Tactile and visual criteria were utilized to validate the clinical efficacy of caries removal in both groups. Moreover, caries removal was confirmed by utilizing caries detector dye (red detector, Cerkamed). Points intensively dyed in red indicated carious dentin. Efficacy was rated and given a numerical value as 0, 1, 2, 3, 4, and 5 according to the Ericson rating scale, as shown in (Table 1).

Table 1 Definition of the scores for caries removal Score Definition 0 Complete removal of caries

1. Caries is found at the cavity floor.
2. Caries is found at the floor and/or one wall.
3. Caries is found at the floor and/ or two walls.
4. Caries is found at the floor and /or more than two walls
5. Caries is found at the margins, walls, and floor of the cavity.

Using impression material and a calibrated insulin syringe for both groups, the amount of removed carious tissue was measured by computing the difference between the cavity's initial volume before caries removal and the final volume of the cavity after caries removal (as previously explained).

All treated cavities were finally restored once all caries had been eliminated.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children of both genders in the age group of 8-11 years and rated as definitely positive or positive using Frankl Behaviour Rating Scale
2. 30 permanent first molars with class I (occlusal) active carious lesion classified as code 5 , according to the international caries detection and assessment system, involving dentin with a cavity opening diameter of 2mm.
3. Permanent molars with absence of peri-apical or inter-radicular radiolucency.

Exclusion Criteria:

1. Molars with developmental anomalies.
2. Decayed molars that show clinical or radiographic evidence of pulpal involvement.
3. Parental refusal to sign the informed consent.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Assessment of caries removal efficiency by visual examination | baseline (immediately after caries removal procedures) Up to 3 minutes, no follow up is required.
  Visual examination to assess the color of dentin and evidence of the presence or absence of soft caries.
Assessment of caries removal efficiency by tactile examination | baseline (immediately after caries removal procedures) Up to 5 minutes, no follow up is required
  Tactile sensation to assess the texture, hardness, and consistency of dentin, i.e.
  the explorer should not stick to the dentin when moved along the surface without a catch or a tug-back sensation.
Assessment of caries removal efficacy by using caries detector dye | baseline (immediately after caries removal procedures) Up to 10 minutes, no follow up is required.
  Caries removal efficacy was assessed using the Ericson rating scale "The Ericson rating scale was used to assess the residual caries. Caries removal status scores are defined as 0, 1,2,3,4, or 5, with 5 indicating the highest residual caries.
Assessment of the volume of the removed carious tissue in cubic millimeters (mm3) | baseline (immediately after caries removal procedures) Up to 15 minutes, no follow up is required.
  Using impression material and a calibrated insulin syringe for both groups, the amount of removed carious tissue was measured by computing the difference between the cavity's initial volume before caries removal and the final volume of the cavity after caries removal

CONTACTS AND LOCATIONS:
Overall Officials: Ghada AH El baz, professor, Principal Investigator — Suez Canal University
Locations (1):
- Faculty of Medicine, Suez canal university, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Yes